CLINICAL TRIAL: NCT05812352
Title: Evaluating Instructional Interventions Supporting Laypeople Addressing Prehospital Hemorrhage Study: A Randomized Controlled Trial
Brief Title: Supporting Laypeople Addressing Prehospital Hemorrhage Study
Acronym: SLAPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Washington University School of Medicine (Other); LFR International (Unknown)
Responsible Party: Principal Investigator, Zachary Eisner, Researcher, University of Michigan
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00229966
Record Dates: First submitted 2023-03-30; First posted 2023-04-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Hemorrhage; Laceration
MeSH Terms: conditions — Hemorrhage; Lacerations

STUDY DESIGN:
Intervention Model Description: Participants are randomized to 1 of 4 educational interventions. Once the initial instructional intervention is completed, participants subsequently present for a 6-month follow-up.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor only enters the laboratory after the participant has attempted to apply the tourniquet. Therefore, the outcomes assessor is unaware of the instructional intervention that was employed. The outcomes assessor will assess (1) tourniquet placement sufficient distance above the injury defined as at least 2 inches proximal to the amputation, (2) turning on an external diaphragm pump that attempts to force water through tubing in the mannequin extremity bypassing the tourniquet.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Audio recording and instructional flashcard with tourniquet ("audio kit") - 6 month follow-up (Experimental): MP3 audio files for each of 6 steps and instructional flashcard with pictures corresponding to each of the 6 steps of tourniquet application, used for tourniquet application attempt. Participants repeat the tourniquet application attempt with the audio kit at 6 month follow-up
  Interventions: Behavioral: Audio kit
- Instructional flashcard with tourniquet - 6 month follow-up (Experimental): Instructional flashcard with pictures corresponding to each of the 6 steps of tourniquet application, used for tourniquet application attempt. Participants repeat the tourniquet application attempt with the instructional flashcard at 6 month follow-up
  Interventions: Behavioral: Instructional flashcard
- In-person training with tourniquet - 6 month follow-up (Experimental): Stop the Bleed bleeding control (B-Con) course is used for instruction for tourniquet application attempt. Participants repeat the tourniquet application attempt without any POC instruction or re-training at 6 month follow-up
  Interventions: Behavioral: In-person training
- Control group with no in-person training and no point-of-care instruction access - 6 month follow-up (No Intervention): There is no in-person training or point-of-care (POC) instructional interventions for this group for tourniquet application attempt. Participants repeat the tourniquet application attempt without any in-person training or POC instructional interventions at 6 month follow-up

INTERVENTIONS:
Behavioral: Audio kit — MP3 audio files for each of 6 steps and instructional flashcard with pictures corresponding to each of the 6 steps of tourniquet application
  Arms: Audio recording and instructional flashcard with tourniquet ("audio kit") - 6 month follow-up
Behavioral: Instructional flashcard — Single page (instructional flashcard) with pictures corresponding to each of the 6 steps of tourniquet application
  Arms: Instructional flashcard with tourniquet - 6 month follow-up
Behavioral: In-person training — Stop the Bleed bleeding control (B-Con) course is used for instruction for tourniquet application attempt
  Arms: In-person training with tourniquet - 6 month follow-up

SUMMARY:
It is unknown if bystanders equipped with point-of-care (POC) instruction are as effective as bystanders with in-person training for bleeding control. Therefore, POC instructional interventions were developed during this study in response to the scalability challenges associated with in-person training to measure the comparative effectiveness and skill retention of POC instructions vs in-person training using a randomized clinical trial design.

DETAILED DESCRIPTION:
Road traffic injuries (RTIs) are the largest contributor to the global trauma burden, which disproportionately affects low- and middle-income countries (LMICs). With a lack of robust emergency medical services (EMS), there has been increasing reliance on layperson bystanders to respond to RTIs in LMICs, called lay first responders (LFRs). In prospective studies of LFR activity across three sub-Saharan African countries comprising 2,039 total patient encounters, LFRs most frequently provided hemorrhage control in 61% of patient encounters. Rapid hemorrhage control for compressible extremity hemorrhage by bystander LFRs has the potential to mitigate exsanguination, reducing mortality secondary to RTIs. Rapid hemorrhage control also has applicability to high-income country settings like the United States that sustain high rates of penetrating trauma due to gun violence. Rapid hemorrhage control using tourniquets for compressible extremity hemorrhage in patients not yet in shock is strongly associated with saved lives demonstrated in battlefield studies, decreasing preventable deaths by more than 50%. Bystanders may be trained in-person or point-of-care (POC) instruction may be provided, as exists with automated external defibrillators. However, it is unknown if bystanders equipped with POC instruction are as effective as bystanders with in-person training for tourniquet application. Therefore, the investigators developed POC instructional interventions in response to the scalability challenges associated with in-person training to measure comparative effectiveness and skill retention using a randomized controlled trial design.

ELIGIBILITY:
Inclusion Criteria:

* Understand spoken and written English

Exclusion Criteria:

* None

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2023-01-24 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Correct tourniquet application at initial encounter | After initial intervention (up to 20 minutes)
  Number of participants who meet all criteria for correct application of the tourniquet
Correct tourniquet application at 6-month follow-up | 6 months
  Number of participants who meet all criteria for correct application of the tourniquet

SECONDARY OUTCOMES:
Level of Participant Confidence initially | After initial intervention (up to 20 minutes)
  Participants will self-rate on a Likert scale of 0 - 10, where 0 is no confidence and 10 is absolutely confident
Level of Participant Confidence at 6-month follow-up | 6 months
  Participants will self-rate on a Likert scale of 0 - 10, where 0 is no confidence and 10 is absolutely confident

CONTACTS AND LOCATIONS:
Overall Officials: Zachary Eisner, BS, Principal Investigator — University of Michigan; Patricia Widder, MS, Study Director — Washington University in St. Louis - McKelvey School of Engineering
Locations (1):
- Washington University in St. Louis - McKelvey School of Engineering, Dept. of Biomedical Engineering, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request to the corresponding author
Supporting Information: Study Protocol
Time Frame: Within 18 months of completion of primary outcome measures